CLINICAL TRIAL: NCT02405780
Title: An Open-label Extension Study to Compare the Long-term Efficacy, Safety, Immunogenicity and Pharmacokinetics of FKB327 and Humira® in Patients With Rheumatoid Arthritis on Concomitant Methotrexate
Brief Title: A Study to Compare FKB327 Long-term Safety, Efficacy and Immunogenicity With Humira® in Rheumatoid Arthritis Patients
Acronym: ARABESC-OLE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fujifilm Kyowa Kirin Biologics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FKB327-003
Record Dates: First submitted 2015-03-17; First posted 2015-04-01 (Estimated); Results first posted 2019-03-26 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Arthritis, Rheumatoid
Keywords: Rheumatoid; Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis | interventions — FKB327; adalimumab biosimilar HS016; Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- FKB327 (Experimental): Patients will receive the drug 40 mg every other week by subcutaneous injection. The treatment period may continue for 76 weeks.
  Interventions: Drug: FKB327
- Humira® (Active Comparator): Patients will receive the drug 40 mg every other week by subcutaneous injection. The treatment period may continue for 76 weeks.
  Interventions: Drug: Humira®

INTERVENTIONS:
Drug: FKB327 — Solution of FKB327 for subcutaneous injection administered in a dose of 40 mg every 2 weeks for 28 weeks. Patients may continue to receive FKB327 40 mg every other week by subcutaneous injection for up to 76 weeks.
  Other Names: adalimumab biosimilar
  Arms: FKB327
Drug: Humira® — Solution of Humira® for subcutaneous injection administered in a dose of 40 mg every 2 weeks for 28 weeks. Patients may then receive FKB327 40 mg every other week by subcutaneous injection from week 30 to week 76.
  Other Names: adalimumab
  Arms: Humira®

SUMMARY:
The purpose of the study is to compare the long-term safety, effectiveness and immunogenicity of FKB327 in comparison to Humira® in rheumatoid arthritis patients who have completed study FKB327-002 and have inadequate disease control on methotrexate.

DETAILED DESCRIPTION:
The first period of this extension study was an open label, randomised, comparative, multi centre, 2 arm extension Phase 3 study in patients with RA who were taking a stable dose of MTX and who had continued from the preceding Study FKB327-002 (NCT02260791). The transition from Study FKB327-002 was ideally to occur without interruption: the Week 24 visit of Study FKB327-002 was to be on the same day as the Week 0 visit of Study FKB327-003. Patients who had received FKB327 in Study FKB327-002 received FKB327 or Humira in a 2:1 ratio and patients who had received Humira in Study FKB327-002 received Humira or FKB327 in a 2:1 ratio (Period I). The second period of the study was an open label, single arm extension in which all patients received FKB327 treatment from Week 30 to Week 76 (Period II), followed by a 4 week Follow up period.

Clinic visits were scheduled for Weeks 0, 2, 4, 8, 12, 24, 30, 32, 34, 42, 54, 66, 76, and 80. The patient or carer was allowed to administer interim doses of study drug at home every other week (eow) between clinic visits.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has completed the Week 24 visit procedures of Study FKB327-002 (NCT02260791) and are continuing with methotrexate
2. In the investigator's opinion, the patient showed a clinical response to treatment during Study FKB327-002 (NCT02260791)

Exclusion Criteria:

1. Patient has evidence of a serious adverse event (SAE) ongoing from Study FKB327-002
2. Patient has presence of active and/or untreated latent tuberculosis (TB)

Other Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 645 (Actual)
Dates: Start 2015-06-10 (Actual); Primary Completion 2018-01-18 (Actual); Study Completion 2018-01-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Josephine Glover, MD, Principal Investigator — Coephycient Pharmaceutical Consultancy
Locations (92):
- United States (15):
  - Research Site, Peoria, Arizona
  - Research Site, Palm Desert, California
  - Research Site, Boca Raton, Florida
  - Research Site, Brandon, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Miami, Florida
  - Research Site, Sarasota, Florida
  - Research Site, Shreveport, Louisiana
  - Research Site, Lansing, Michigan
  - Research Site, Durham, North Carolina
  - Research Site, Middleburg Heights, Ohio
  - Research Site, Duncansville, Pennsylvania
  - Research Site, Amarillo, Texas
  - Research Site, Austin, Texas
  - Research Site, Mesquite, Texas
- Canada (2):
  - Research Site, Saint Catherines, Ontario
  - Research Site, Trois-Rivières, Quebec
- Chile (5):
  - Research Site, Osorno
  - Research Site, Puerto Varas
  - Research Site G, Santiago
  - Research Site M, Santiago
  - Research Site, Temuco
- Czechia (6):
  - Research Site, Brno
  - Research Site, Hlučín
  - Research Site U, Prague
  - Research Site, Prague
  - Research Site, Uherské Hradiště
  - Research Site, Zlín
- Germany (5):
  - Research Site, Aachen
  - Research Site, Berlin
  - Research Site, Hamburg
  - Research Site, Munich
  - Research Site, Ratingen
- Peru (6):
  - Research Site B, Arequipa
  - Research Site M, Arequipa
  - Research Site CA, Lima
  - Research Site CH, Lima
  - Research Site PA, Lima
  - Research Site S, Lima
- Poland (10):
  - Research Site D, Bialystok
  - Research Site R, Bialystok
  - Research Site, Gdynia
  - Research Site, Katowice
  - Research Site KL, Krakow
  - Research Site KR, Krakow
  - Research Site, Lublin
  - Research Site P, Poznan
  - Research Site RH, Poznan
  - Research Site, Torun
- Romania (8):
  - Research Site, Oradea, Bihor County
  - Research Site, Sfântu Gheorghe, Covasna
  - Research Site, Brasov
  - Research Site, Brăila
  - Research Site C, Bucharest
  - Research Site R, Bucharest
  - Research Site T, Bucharest
  - Research Site, Galati
- Russia (17):
  - Research Site, Ufa, Bashkortostan Republic
  - Research Site, Petrozavodsk, Karelia Republic
  - Research Site, Kazan', Tatarstan Republic
  - Research Site D, Moscow
  - Research Site SM, Moscow
  - Research Site ST, Moscow
  - Research Site, Nizhny Novgorod
  - Research Site, Penza
  - Research Site, Perm
  - Research Site, Ryazan
  - Research Site B, Saint Petersburg
  - Research Site Z, Saint Petersburg
  - Research Site, Saratov
  - Research Site, Smolensk
  - Research Site, Vladimir
  - Research Site E, Yaroslavl
  - Research Site S, Yaroslavl
- Spain (4):
  - Research Site, Santiago de Compostela, La Coruna
  - Research Site, Bilbao, Vizcaya
  - Research Site G, Barcelona
  - Research Site, Málaga
- Ukraine (14):
  - Research Site, Chernivtsi
  - Research Site, Ivano-Frankivsk
  - Research Site A, Kyiv
  - Research Site B, Kyiv
  - Research Site P, Kyiv
  - Research Site, Lutsk
  - Research Site C, Lviv
  - Research Site N, Lviv
  - Research Site, Poltava
  - Research Site, Ternopil
  - Research Site, Uzhhorod
  - Research Site G, Vinnytsia
  - Research Site Sh, Vinnytsia
  - Research Site St, Vinnytsia

REFERENCES:
- [Derived] Huizinga TWJ, Torii Y, Muniz R. Adalimumab Biosimilars in the Treatment of Rheumatoid Arthritis: A Systematic Review of the Evidence for Biosimilarity. Rheumatol Ther. 2021 Mar;8(1):41-61. doi: 10.1007/s40744-020-00259-8. Epub 2020 Dec 1. PMID 33263165
- [Derived] Genovese MC, Glover J, Greenwald M, Porawska W, El Khouri EC, Dokoupilova E, Vargas JI, Stanislavchuk M, Kellner H, Baranova E, Matsunaga N, Alten R. FKB327, an adalimumab biosimilar, versus the reference product: results of a randomized, Phase III, double-blind study, and its open-label extension. Arthritis Res Ther. 2019 Dec 12;21(1):281. doi: 10.1186/s13075-019-2046-0. PMID 31831079

RESULTS

PARTICIPANT FLOW:
Groups:
- FKB327-FKB327-FKB327: Period I: This is the treatment arm where subjects had been treated with FKB327 in the preceding study, FKB327-002 and were re-randomized to FKB327 in Period I of study FKB327-003 (F-F).
  Period II: From week 30 all subjects received FKB327; (F-F-F).
- FKB327-Humira-FKB327: Period I: This is the treatment arm where subjects had been treated with FKB327 in the preceding study FKB327-002 and were re-randomized to the reference product, Humira, during Period I of study FKB327-003 (F-H).
  Period II: From week 30 all subjects received FKB327; (F-H-F).
- Humira-FKB327-FKB327: Period I: This is the treatment arm where subjects had been treated with the reference product Humira in the preceding study, FKB327-002 and were re-randomized to FKB327 during Period I of study FKB327-003 (H-F).
  Period II: From week 30 all subjects received FKB327; (H-F-F).
- Humira-Humira-FKB327: Period I: This is the treatment arm where subjects had been treated with the reference product Humira in the preceding study, FKB327-002, and were re-randomized to the reference product Humira during Period I of study FKB327-003 (H-H).
  Period II: From week 30 all subjects received FKB327; (H-H-F).
Period: Period I
Arm/Group | FKB327-FKB327-FKB327 | FKB327-Humira-FKB327 | Humira-FKB327-FKB327 | Humira-Humira-FKB327
Started | 216 | 108 | 108 | 213
Completed | 189 | 100 | 93 | 190
Not Completed | 27 | 8 | 15 | 23
Not completed — Adverse Event | 8 | 0 | 3 | 7
Not completed — Medical reasons | 1 | 1 | 0 | 1
Not completed — Screening Failure | 1 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 9 | 1 | 3 | 4
Not completed — Non-compliance with study procedures | 8 | 6 | 8 | 11
Period: Period II
Arm/Group | FKB327-FKB327-FKB327 | FKB327-Humira-FKB327 | Humira-FKB327-FKB327 | Humira-Humira-FKB327
Started | 189 | 100 | 93 | 190
Completed | 174 | 88 | 81 | 172
Not Completed | 15 | 12 | 12 | 18
Not completed — Adverse Event | 3 | 5 | 4 | 11
Not completed — Medical reason | 0 | 1 | 0 | 0
Not completed — Pregnancy | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 7 | 4 | 0 | 3
Not completed — Non-compliance with study procedures | 5 | 2 | 7 | 4

BASELINE CHARACTERISTICS:
Groups:
- FKB327-FKB327: This is the treatment arm where subjects had been treated with FKB327 in the preceding study, FKB327-002 and were re-randomized to receive FKB327 in Study FKB327-003.
- FKB327-Humira: This is the treatment arm where subjects had been treated with FKB327 in the preceding study, FKB327-002 and were re-randomized to receive the reference product Humira in Study FKB327-003.
- Humira-FKB327: This is the treatment arm where subjects had been treated with the reference product Humira in the preceding study, FKB327-002 and were re-randomized to receive FKB327 in Study FKB327-003.
- Humira-Humira: This is the treatment arm where subjects had been treated with the reference product Humira in the preceding study, FKB327-002 and were re-randomized to receive the reference product Humira in Study FKB327-003.
- Total: Total of all reporting groups
Arm/Group | FKB327-FKB327 | FKB327-Humira | Humira-FKB327 | Humira-Humira | Total
Number analyzed (Participants) | 216 | 108 | 108 | 213 | 645
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 183 | 92 | 96 | 169 | 540
  >=65 years | 33 | 16 | 12 | 44 | 105
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 162 | 85 | 83 | 171 | 501
  Male | 54 | 23 | 25 | 42 | 144
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1 | 2
  Asian | 1 | 0 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 2 | 2 | 6
  White | 187 | 90 | 90 | 185 | 552
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 26 | 17 | 15 | 25 | 83
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 1 | 1 | 1 | 2 | 5
  Chile | 13 | 7 | 6 | 14 | 40
  Czechia | 22 | 9 | 11 | 22 | 64
  Germany | 7 | 4 | 3 | 8 | 22
  Peru | 26 | 17 | 15 | 26 | 84
  Poland | 41 | 22 | 22 | 39 | 124
  Romania | 8 | 4 | 3 | 8 | 23
  Russia | 33 | 18 | 16 | 29 | 96
  Spain | 2 | 1 | 2 | 4 | 9
  Ukraine | 39 | 14 | 17 | 37 | 107
  United States | 24 | 11 | 12 | 24 | 71

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Adverse Events as a Measure of Safety Per Treatment Group in Period I
Description: Period I: Patients were carefully monitor for Adverse Events from signing of informed consent until week 30 and thereafter during Period II of the study. For patients who discontinued early, a follow-up period of 4 weeks was added to the Early Termination Visit.
  The investigator actively asked the patients for Adverse Events. Patients spontaneously reported Adverse Events to the Investigator during clinic visits or in between visits.
Time Frame: Period I: from Week 0 up until Week 30;
Population: Each patient was counted once within each System Organ Class (SOC) and Preferred Term (PT). A patient may have had multiple events counted. Treatment Emergen Adverse Events (TEAE) defined as AEs that started or increased in severity after the first study dose and counted under the treatment arm.
Measure: Number; unit: participants
Groups:
- FKB327-FKB327: Period I: This is the treatment arm where subjects had been treated with FKB327 in the preceding study, FKB327-002 and were re-randomized to FKB327 in Period I of study FKB327-003 (F-F).
- FKB327-Humira: Period I: This is the treatment arm where subjects had been treated with FKB327 in the preceding study FKB327-002 and were re-randomized to the reference product, Humira, during Period I of study FKB327-003 (F-H).
- Humira-FKB327: Period I: This is the treatment arm where subjects had been treated with the reference product Humira in the preceding study, FKB327-002 and were re-randomized to FKB327 during Period I of study FKB327-003 (H-F).
- Humira-Humira: Period I: This is the treatment arm where subjects had been treated with the reference product Humira in the preceding study, FKB327-002, and were re-randomized to the reference product Humira during Period I of study FKB327-003 (H-H).
Arm/Group | FKB327-FKB327 | FKB327-Humira | Humira-FKB327 | Humira-Humira
Number analyzed (Participants) | 216 | 108 | 108 | 213
participants
  Death | 0 | 0 | 1 | 1
  Treatment Emergent Deaths | 0 | 0 | 1 | 1
  At least 1 TEAE | 103 | 59 | 59 | 117
  At least 1 severe TEAE | 5 | 2 | 3 | 2
  At least 1 treatment related TEAE | 39 | 21 | 27 | 49
  Premature Discontinuation due to a TEAE | 10 | 0 | 4 | 11
  Treatment Interruption due to a TEAE | 19 | 9 | 14 | 20

2. Primary Outcome: Number of Patients With Adverse Events as a Measure of Safety in Period II - Single Treatment Period
Description: From week 30 all subjects were transferred to receive FKB327 treatment. Adverse Events were contentiously monitored and recorded during Period II. For patients discontinuing the study prematurely, a follow-up period of 4 weeks was added to the Early Termination Visit. The data for Period II is based on the number of patients in the Safety Analysis Set that entered Period II.
Time Frame: Period II: from Week 30 up to Week 80
Measure: Count of Participants; unit: Participants
Groups:
- FKB327: Period II: From week 30 all patients received one subcutaneous injection every other week of 40 mg/0.8 mL presented in an auto-injector (AI) or in a pre-filled syringe (PFS).
  Based on the design of the study and to what treatment groups the subjects were randomised to in Period I, some patients received continuous treatment with FKB327 40 mg/0.8mL every other week by subcutaneous injection for up to 76 weeks. This was applicable to subjects in treatment groups (F-F-F) and (H-F-F)
Arm/Group | FKB327
Number analyzed (Participants) | 572
Participants
  Death | 2
  Treatment Emergent Deaths | 2
  At least 1 TEAE | 340
  At least 1 severe TEAE | 19
  At least 1 treatment related TEAE | 126
  Premature Discontinuation due to a TEAE | 25
  Treatment Interruption due to a TEAE | 36

3. Primary Outcome: Number of Patients With Serious Adverse Events as a Measure of Safety Per Treatment Group in Period I
Description: A Serious Adverse Event (SAE) was defined in the Protocol as: Death; or a Life-threatening Adverse Event (AE); Inpatient Hospitalization; Persistant or significant disability or incapacity; A congenital anomaly/birth defect; An important medical event that may not have resulted in death, have been life-threatening, or required hospitalization, but may have jeopardized the patient and may have required medical intervention to prevent 1 of the outcomes listed in this definition.
  SAEs were followed until resolution, the investigator confirmed the event was unlikely to resolve or the patient was recorded as lost to follow-up.
Time Frame: Period I: from Week 0 up until Week 30
Population: Each patient was counted once within each System Organ Class (SOC) and Preferred Term (PT). Death defined as a fatal outcome of a (S) AE.
Measure: Number; unit: participants
Arm/Group | FKB327-FKB327 | FKB327-Humira | Humira-FKB327 | Humira-Humira
Number analyzed (Participants) | 216 | 108 | 108 | 213
participants
  Deaths | 0 | 0 | 1 | 1
  Treatment Emergent Deaths | 0 | 0 | 1 | 1
  Treatment Discontinuation due to a TESAE | 0 | 0 | 0 | 2
  Treatment Interruption due to a TESAE | 3 | 2 | 4 | 2
  At least 1 TESAE | 5 | 7 | 5 | 7
  Number of TESAE | 7 | 9 | 9 | 7
  At least 1 SAE | 5 | 7 | 5 | 7

4. Primary Outcome: Number of Patients With Serious Adverse Events as a Measure of Safety in Period II - Single Treatment Period
Description: Period II: at week 30 all patients were transferred to receive FKB327.
  Each subject was counted once within each System Organ Class (SOC) and Preferred Term (PT). Death defined as a fatal outcome of a (S)AE.
  SAEs were followed until resolution, the investigator confirmed the event was unlikely to resolve or the patient was lost to follow-up.
Time Frame: Period II: from Week 30 up to Week 80
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Groups:
- FKB327: Period II: From week 30 all subjects received one subcutaneous injection every other week of FKB327 40 mg/0.8 mL presented in an auto-injector (AI) or in a pre-filled syringe (PFS) .
  Based on the design of the study and to what treatment groups the subjects were randomised to in Period I, some patients received continuous treatment with FKB327 40 mg/0.8mL every other week by subcutaneous injection for up to 76 weeks. This was applicable to subjects in treatment groups (F-F-F) and (H-F-F)
Arm/Group | FKB327
Number analyzed (Participants) | 572
Participants
  Death | 2
  Treatment Emergent Deaths | 2
  At least 1 severe TEAE | 19
  Treatment Discontinuation due to a TESEA | 10
  Treatment Interruption due to a TESAE | 6
  At least 1 TESAE | 33
  Number of TESAE | 45
  At least 1 SAE | 33

5. Primary Outcome: Changes in Vital Signs as a Measure of Safety - Systolic Blood Pressure
Description: Systolic Blood Pressure is part of Vital Signs which were part of the subject safety evaluations. Systolic Blood Pressure was measured at the following time-points: Week 0, Week 4, Week 8, Week 12, Week 24 and Week 80/End o Study (EOS). Systolic Blood Pressure with changes from Baseline_002 (NCT022600791) was summarized by treatment sequence over the whole study period for each visit.
  Baseline_002 is defined as the last non-missing measurement collected prior to the first study medication administered at Week 0 from Study FKB327-002.
Time Frame: From Week 0 to Week 80
Population: The number of patients in the Safety Analysis Set; is equal to the number of patients who entered Period I. The number of patients at the following visit is the number of patients who at a given timepoint had a measurement completed for the Safety Analysis Set.
Measure: Median (Full Range); unit: mmHg
Groups:
- FKB327-FKB327-FKB327: Period I: This is the treatment arm where subjects had been treated with FKB327 in the preceding study, FKB327-002 and were re-randomized to receive FKB327 in Study FKB327-003 (F-F).
  Period II: From week 30 all subjects received FKB327 (F-F-F).
- FKB327-Humira-FKB327: Period I: This is the treatment arm where subjects had been treated with FKB327 in the preceding study, FKB327-002 and were re-randomized to receive the reference product Humira in Study FKB327-003 (F-H).
  Period II: From week 30 all subjects received FKB327 (F-H-F).
- Humira-FKB327-FKB327: Period I: This is the treatment arm where subjects had been treated with the reference product Humira in the preceding study, FKB327-002 and were re-randomized to receive FKB327 in Study FKB327-003 (H-F).
  Period II: From week 30 all subjects received FKB327 (H-F-F).
- Humira-Humira-FKB327: Period I: This is the treatment arm where subjects had been treated with the reference product Humira in the preceding study, FKB327-002 and were re-randomized to receive the reference product Humira in Study FKB327-003 (H-H).
  Period II: From week 30 all subjects received FKB327 (H-H-F).
Arm/Group | FKB327-FKB327-FKB327 | FKB327-Humira-FKB327 | Humira-FKB327-FKB327 | Humira-Humira-FKB327
Number analyzed (Participants) | 216 | 108 | 108 | 213
mmHg
  Baseline_002 | 125.0 [86 to 168] | 125.5 [94 to 174] | 131.0 [88 to 167] | 129.0 [90 to 162]
  Week 0 | 125.0 [84 to 166] | 123.5 [90 to 160] | 127.0 [98 to 179] | 125.0 [90 to 163]
  Changes from Baseline_002 at week 0 | 0.0 [-34 to 35] | -2.0 [-30 to 32] | -2.0 [-44 to 32] | -2.0 [-50 to 51]
  Week 4: number analyzed (Participants) | 213 | 106 | 107 | 208
  Week 4 | 124.0 [82 to 172] | 125.0 [95 to 164] | 124.0 [92 to 186] | 125 [94 to 167]
  Changes from Baseline_002 at week 4: number analyzed (Participants) | 213 | 106 | 107 | 208
  Changes from Baseline_002 at week 4 | 0.0 [-56 to 38] | 0.0 [-22 to 44] | -6.0 [-39 to 39] | -1.0 [-37 to 36]
  Week 8: number analyzed (Participants) | 205 | 104 | 104 | 204
  Week 8 | 124.0 [88 to 154] | 124.0 [89 to 153] | 128.0 [92 to 160] | 125.0 [92 to 156]
  Changes from Baseline_002 at week 8: number analyzed (Participants) | 205 | 104 | 104 | 204
  Changes from Baseline_002 at week 8 | -2.0 [-47 to 32] | -0.5 [-28 to 41] | -1.5 [-35 to 30] | -2.0 [-38 to 36]
  Week 12: number analyzed (Participants) | 204 | 104 | 103 | 204
  Week 12 | 125.0 [91 to 159] | 124.5 [86 to 165] | 126.0 [89 to 167] | 125.0 [92 to 170]
  Changes from Baseline_002 at week 12: number analyzed (Participants) | 204 | 104 | 103 | 204
  Changes from Baseline_002 at week 12 | 0.0 [-35 to 45] | -2.0 [-40 to 35] | -2.0 [-44 to 28] | 0.0 [-46 to 40]
  Week 24: number analyzed (Participants) | 198 | 102 | 97 | 200
  Week 24 | 125.0 [90 to 155] | 127.5 [92 to 156] | 125.0 [86 to 163] | 126.0 [94 to 176]
  Changes from Baseline_002 at week 24: number analyzed (Participants) | 198 | 102 | 97 | 200
  Changes from Baseline_002 at week 24 | -2.0 [-46 to 36] | 0.0 [-38 to 33] | -5.0 [-44 to 28] | 0.0 [-49 to 37]
  Week 80/EOS: number analyzed (Participants) | 174 | 88 | 81 | 172
  Week 80/EOS | 126.0 [90 to 157] | 125.0 [88 to 171] | 126.0 [91 to 163] | 125.0 [98 to 163]
  Changes from Baseline_002 at week 80/EOS: number analyzed (Participants) | 174 | 88 | 81 | 172
  Changes from Baseline_002 at week 80/EOS | -0.5 [-53 to 53] | 0.0 [-37 to 41] | -2.0 [-47 to 27] | -1.5 [-42 to 26]

6. Primary Outcome: Changes in Vital Signs as a Measure of Safety - Diastolic Blood Pressure
Description: Diastolic Blood Pressure is part of Vital Signs which were part of the subject safety evaluations. Diastolic Blood Pressure was measured at the following time-points: Week 0, Week 4, Week 8, Week 12, Week 24 and Week 80/End o Study (EOS). Diastolic Blood Pressure with changes from Baseline_002 (NCT022600791) was summarized by treatment sequence over the whole study period for each visit measured.
  Baseline_002 is defined as the last non-missing measurement collected prior to the first study medication administered at Week 0 from Study FKB327-002.
Time Frame: From Week 0 to Week 80
Population: as for outcome 5
Measure: Median (Full Range); unit: mmHg
Arm/Group | FKB327-FKB327-FKB327 | FKB327-Humira-FKB327 | Humira-FKB327-FKB327 | Humira-Humira-FKB327
Number analyzed (Participants) | 216 | 108 | 108 | 213
mmHg
  Baseline_002 | 78.0 [48 to 99] | 78.0 [56 to 98] | 80.0 [54 to 96] | 77.0 [55 to 105]
  Week 0 | 78.0 [49 to 94] | 75.0 [53 to 102] | 77.0 [57 to 108] | 76.0 [50 to 99]
  Changes from Baseline_002 at week 0 | 0.0 [-23 to 28] | -1.5 [-25 to 22] | -1.0 [-25 to 24] | 0.0 [-31 to 23]
  Week 4: number analyzed (Participants) | 213 | 106 | 107 | 208
  Week 4 | 76.0 [51 to 94] | 77.0 [59 to 96] | 76.0 [58 to 107] | 78.0 [55 to 100]
  Changes from Baseline_002 at week 4: number analyzed (Participants) | 213 | 106 | 107 | 208
  Changes from Baseline_002 at week 4 | 0.0 [-33 to 28] | 0.0 [-18 to 36] | 0.0 [-22 to 25] | 0.0 [-27 to 30]
  Week 8: number analyzed (Participants) | 205 | 104 | 104 | 204
  Week 8 | 78.0 [59 to 97] | 78.0 [58 to 99] | 80.0 [57 to 97] | 77.0 [51 to 95]
  Changes from Baseline_002 at week 8: number analyzed (Participants) | 205 | 104 | 104 | 204
  Changes from Baseline_002 at week 8 | 0.0 [-26 to 26] | 0.0 [-23 to 34] | 0.0 [-18 to 15] | 0.0 [-30 to 21]
  Week 12: number analyzed (Participants) | 204 | 104 | 103 | 204
  Week 12 | 78.0 [52 to 98] | 78.5 [56 to 104] | 80.0 [58 to 103] | 78.0 [58 to 95]
  Changes from Baseline_002 at week 12: number analyzed (Participants) | 204 | 104 | 103 | 204
  Changes from Baseline_002 at week 12 | 0.0 [-26 to 23] | 0.0 [-24 to 21] | 0.0 [-15 to 31] | 0.0 [-26 to 20]
  Week 24: number analyzed (Participants) | 198 | 102 | 97 | 200
  Week 24 | 78.0 [52 to 96] | 78.0 [52 to 99] | 78.0 [50 to 104] | 78.0 [55 to 96]
  Changes from Baseline_002 at week 24: number analyzed (Participants) | 198 | 102 | 97 | 200
  Changes from Baseline_002 at week 24 | 1.0 [-22 to 25] | 0.0 [-24 to 19] | 0.0 [-22 to 16] | 0.0 [-36 to 18]
  Week 80/EOS: number analyzed (Participants) | 174 | 88 | 81 | 172
  Week 80/EOS | 78.0 [41 to 98] | 79.0 [60 to 100] | 80.0 [56 to 102] | 77.0 [50 to 95]
  Changes from Baseline_002 at week 80/EOS: number analyzed (Participants) | 174 | 88 | 81 | 172
  Changes from Baseline_002 at week 80/EOS | 0.0 [-42 to 30] | 0.0 [-32 to 24] | 0.0 [-25 to 18] | 0.0 [-48 to 20]

7. Primary Outcome: Changes in Vital Signs as a Measure of Safety - Pulse Rate
Description: Pulse rate is part of Vital Signs which were part of the subject safety evaluations. Pulse rate was measured at the following time-points: Weeks 0, 4, 8, 12, 24 and 80/End of Study (EOS). Pulse Rate with changes from Baseline_002 (NCT022600791) was summarized by treatment sequence over the whole study period for each visit.
  Baseline_002 is defined as the last non-missing measurement collected prior to the first study medication administered at Week 0 from Study FKB327-002.
Time Frame: From Week 0 to Week 80
Population: The number of patients in the Safety Analysis Set; is equal to the number of patients who entered Period I. The number of patients at the following visits is the number of patients who at a given time point had a measurement completed for the Safety Analysis Set.
Measure: Median (Full Range); unit: Beats per minute (bpm)
Arm/Group | FKB327-FKB327-FKB327 | FKB327-Humira-FKB327 | Humira-FKB327-FKB327 | Humira-Humira-FKB327
Number analyzed (Participants) | 216 | 108 | 108 | 213
Beats per minute (bpm)
  Baseline_002 | 74.0 [51 to 100] | 74.0 [54 to 97] | 74.0 [54 to 102] | 74.0 [53 to 106]
  Week 0 | 72.0 [50 to 102] | 71.0 [48 to 94] | 72.0 [53 to 110] | 72.0 [42 to 99]
  Changes from Baseline_002 at week 0 | -0.5 [-32 to 28] | -3.0 [-28 to 24] | -3.0 [-23 to 44] | -2.0 [-36 to 29]
  Week 4: number analyzed (Participants) | 213 | 106 | 107 | 208
  Week 4 | 72.0 [47 to 112] | 72.0 [52 to 94] | 74.0 [51 to 105] | 72.0 [50 to 102]
  Changes from Baseline_002 at week 4: number analyzed (Participants) | 213 | 106 | 107 | 208
  Changes from Baseline_002 at week 4 | -2.0 [-29 to 24] | -2.0 [-28 to 24] | -2.0 [-24 to 30] | -1.0 [-37 to 32]
  Week 8: number analyzed (Participants) | 205 | 104 | 104 | 204
  Week 8 | 72.0 [53 to 99] | 72.0 [54 to 102] | 72.0 [53 to 100] | 72 [46 to 99]
  Changes from Baseline_002 at week 8: number analyzed (Participants) | 205 | 104 | 104 | 204
  Changes from Baseline_002 at week 8 | 0.0 [-41 to 26] | -2.0 [-26 to 32] | -2.0 [-28 to 19] | -2.0 [-37 to 25]
  Week 12: number analyzed (Participants) | 204 | 104 | 103 | 204
  Week 12 | 71.0 [50 to 98] | 72.0 [56 to 100] | 72.0 [57 to 97] | 71.0 [52 to 92]
  Changes from Baseline_002 at week 12: number analyzed (Participants) | 204 | 104 | 103 | 204
  Changes from Baseline_002 at week 12 | -2.0 [-36 to 30] | -1.5 [-31 to 18] | -1.0 [-28 to 25] | -2.0 [-30 to 19]
  Week 24: number analyzed (Participants) | 198 | 102 | 97 | 200
  Week 24 | 73.0 [50 to 103] | 72.0 [55 to 96] | 72.0 [58 to 99] | 72.0 [49 to 95]
  Changes from Baseline_002 at week 24: number analyzed (Participants) | 198 | 102 | 97 | 200
  Changes from Baseline_002 at week 24 | 0.0 [-35 to 26] | -2.0 [-33 to 20] | -2.0 [-29 to 26] | -2.0 [-32 to 34]
  Week 80/EOS: number analyzed (Participants) | 174 | 88 | 81 | 172
  Week 80/EOS | 74.0 [52 to 110] | 72.0 [55 to 94] | 72.0 [50 to 96] | 73.5 [45 to 111]
  Changes from Baseline_002 at week 80/EOS: number analyzed (Participants) | 174 | 88 | 81 | 172
  Changes from Baseline_002 at week 80/EOS | -1.0 [-31 to 32] | -2.0 [-30 to 19] | -1.0 [-25 to 26] | -1.0 [-37 to 31]

8. Primary Outcome: Changes in Vital Signs as a Measure of Safety - Temperature Measurements
Description: Temperature measurements forms part of the vital signs which was one of the continuous safety measurements for the study primary endpoint.
  Temperature was measured at week 0, week 4, week 8, week 12, week 24 and at week 80 or at End of Study (EOS).
  Temperature with change from Baseline_002 were summarized by treatment sequence over the whole study period.
  Baseline_002 is defined as the last non-missing measurement collected prior to the first study medication administration at Week 0 from Study FKB327-002 (NCT02260791).
Time Frame: From Week 0 to Week 80
Population: The number of patients in the Safety Analysis Set; is equal to the number of patients who entered Period I. The number of patients at the following visits is the number of patients who at a given timepoint had a measurement completed for the Safety Analysis Set.
Measure: Median (Full Range); unit: Centigrades
Arm/Group | FKB327-FKB327-FKB327 | FKB327-Humira-FKB327 | Humira-FKB327-FKB327 | Humira-Humira-FKB327
Number analyzed (Participants) | 216 | 108 | 108 | 213
Centigrades
  Baseline_002 | 36.600 [35.61 to 37.20] | 36.600 [35.50 to 37.00] | 36.600 [35.60 to 37.30] | 36.500 [35.60 to 37.60]
  Week 0 | 36.500 [35.70 to 37.20] | 36.500 [35.50 to 37.10] | 36.600 [35.56 to 37.20] | 36.500 [35.70 to 37.10]
  Changes from Baseline_002 at week 0 | 0.000 [-0.80 to 1.19] | 0.000 [-1.20 to 0.70] | 0.000 [-0.70 to 1.00] | 0.000 [-1.00 to 0.80]
  Week 4: number analyzed (Participants) | 213 | 106 | 107 | 208
  Week 4 | 36.500 [34.56 to 37.70] | 36.500 [35.70 to 37.00] | 36.500 [35.20 to 37.11] | 36.500 [35.60 to 37.20]
  Changes from Baseline_002 at week 4: number analyzed (Participants) | 213 | 106 | 107 | 208
  Changes from Baseline_002 at week 4 | 0.000 [-1.94 to 1.40] | 0.000 [-0.70 to 1.20] | -0.100 [-1.20 to 1.00] | 0.000 [-1.20 to 1.00]
  Week 8: number analyzed (Participants) | 205 | 104 | 104 | 204
  Week 8 | 36.500 [35.00 to 37.28] | 36.500 [35.40 to 37.20] | 36.500 [35.60 to 37.20] | 36.500 [35.50 to 37.30]
  Changes from Baseline_002 at week 8: number analyzed (Participants) | 205 | 104 | 104 | 204
  Changes from Baseline_002 at week 8 | 0.000 [-1.50 to 1.19] | -0.100 [-0.83 to 1.10] | -0.025 [-0.70 to 0.80] | 0.000 [-1.40 to 1.20]
  Week 12: number analyzed (Participants) | 204 | 104 | 103 | 204
  Week 12 | 36.500 [35.56 to 37.20] | 36.500 [35.10 to 37.10] | 36.500 [35.40 to 37.00] | 36.500 [35.60 to 37.40]
  Changes from Baseline_002 at week 12: number analyzed (Participants) | 204 | 104 | 103 | 204
  Changes from Baseline_002 at week 12 | 0.000 [-0.94 to 0.80] | 0.000 [-1.10 to 0.80] | -0.100 [-1.10 to 0.90] | 0.000 [-1.60 to 1.30]
  Week 24: number analyzed (Participants) | 198 | 102 | 97 | 200
  Week 24 | 36.500 [35.50 to 37.20] | 36.500 [35.50 to 37.90] | 36.500 [35.60 to 37.40] | 36.500 [35.60 to 37.20]
  Changes from Baseline_002 at week 24: number analyzed (Participants) | 198 | 102 | 97 | 200
  Changes from Baseline_002 at week 24 | 0.000 [-1.00 to 1.00] | 0.000 [-0.90 to 1.40] | 0.000 [-0.90 to 1.00] | 0.000 [-1.10 to 0.80]
  Week 80/EOS: number analyzed (Participants) | 174 | 88 | 81 | 172
  Week 80/EOS | 36.500 [35.60 to 37.30] | 36.500 [35.70 to 37.10] | 36.500 [35.30 to 37.00] | 36.500 [35.50 to 37.30]
  Changes from Baseline_002 at week 80/EOS: number analyzed (Participants) | 174 | 88 | 81 | 172
  Changes from Baseline_002 at week 80/EOS | 0.000 [-1.10 to 1.19] | 0.000 [-0.80 to 0.90] | -0.100 [-1.00 to 0.70] | 0.000 [-1.00 to 0.90]

9. Primary Outcome: Summary of Most Common Clinical Significant Laboratory Parameters Reported as Adverse Events (Reported by ≥1% of the Patients)
Description: Clinical Laboratory tests for hematology and serum chemistry were performed by the sites and analysed at a Central Laboratory. Urine dip-stick tests were performed by the sites. Laboratory samples were taken at the following time-points (weeks): 0; 4; 8; 12; 24; 30; 42; 54; 66; 76 and 80/End of Study (EOS). Each result outside its normal range was review and assessed by the investigator whether or not it was Clinically Significant (CS) or Not Clinically Significant (NCS) CS laboratory abnormalities were recorded as AEs.
Time Frame: From Week 0 to Week 80
Measure: Number; unit: participants
Groups:
- FKB327-FKB327: Period I: This is the treatment arm where subjects had been treated with FKB327 in the preceding study, FKB327-002 and were re-randomized to receive FKB327 in Study FKB327-003 (F-F).
- FKB327-Humira: Period I: This is the treatment arm where subjects had been treated with FKB327 in the preceding study, FKB327-002 and were re-randomized to receive the reference product Humira in Study FKB327-003 (F-H).
- Humira-FKB327: Period I: This is the treatment arm where subjects had been treated with the reference product Humira in the preceding study, FKB327-002 and were re-randomized to receive FKB327 in Study FKB327-003 (H-F).
- Humira-Humira: Period I: This is the treatment arm where subjects had been treated with the reference product Humira in the preceding study, FKB327-002 and were re-randomized to receive the reference product Humira in Study FKB327-003 (H-H).
- FKB327 Period II: From Week 30 all patients were treated with FKB327
Arm/Group | FKB327-FKB327 | FKB327-Humira | Humira-FKB327 | Humira-Humira | FKB327 Period II
Number analyzed (Participants) | 216 | 108 | 108 | 213 | 572
participants
  Anaemia | 3 | 1 | 2 | 3 | 11
  Leukopenia | 3 | 1 | 0 | 0 | 2
  Neutropenia | 3 | 0 | 0 | 1 | 2
  ALT increased | 3 | 2 | 0 | 1 | 10
  AST increased | 3 | 0 | 0 | 1 | 7
  Dyslipidaemia | 1 | 0 | 1 | 1 | 8
  Hypercholesterolaemia | 3 | 3 | 2 | 3 | 2
  CRP increased | 0 | 0 | 0 | 1 | 8
  Latent TB | 3 | 0 | 4 | 4 | 10
  Mycobacterium tuberculosis complex test positive | 7 | 2 | 2 | 6 | 5
  Haematuria | 1 | 0 | 2 | 2 | 2

10. Secondary Outcome: Changes in Disease Activity Score 28 Based on C Reactive Protein (DAS28 CRP) Score Compared to Baseline as a Measure of Efficacy
Description: The DAS28 score is a combined index that has been developed to measure the disease activity in patients with Rheumatoid arthritis (RA) and has been extensively validated for the use in clinical studies. The DAS28-CRP assessment involved evaluating the number of tender (TJC) and the swollen (SJC) joints (out of 28 specified joints), serum CRP, and patient global assessment of disease activity (Visual analogue scale (VAS) from 0-100, very well to extremely bad). The individual results are summarized using a formula. DAS28 is a number on a scale from 0 to 10 indicating the current activity of the patient's RA. A higher score indicates higher disease activity.
  During the FKB327-003 study for Period I and Period II the DAS28-CRP score was compared to Baseline in study FKB327-002 (NCT02260791).
Time Frame: From Week 0 of FKB327-002 to Week 80
Population: DAS28-CRP and change from Baseline in Study FKB327-002 (i.e. Baseline_002) in DAS28-CRP were summarized by overall treatment sequence and visit as well as by treatment for each period (Period I and Period II)
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | FKB327-FKB327-FKB327 | FKB327-Humira-FKB327 | Humira-FKB327-FKB327 | Humira-Humira-FKB327
Number analyzed (Participants) | 216 | 108 | 108 | 213
units on a scale
  Baseline_002: number analyzed (Participants) | 215 | 107 | 108 | 213
  Baseline_002 | 6.02 [3.3 to 8.1] | 6.12 [2.9 to 8.5] | 5.99 [3.7 to 7.9] | 6.11 [4.0 to 8.0]
  Week 0: number analyzed (Participants) | 215 | 108 | 108 | 213
  Week 0 | 3.46 [1.2 to 7.3] | 3.49 [1.2 to 7.4] | 3.65 [1.2 to 7.2] | 3.36 [1.2 to 7.0]
  Week 0 change from Baseline: number analyzed (Participants) | 214 | 107 | 108 | 213
  Week 0 change from Baseline | -2.56 [-5.7 to 1.0] | -2.63 [-6.4 to 1.2] | -2.33 [-5.4 to 0.9] | -2.75 [-5.7 to 1.3]
  Week 4: number analyzed (Participants) | 208 | 104 | 105 | 203
  Week 4 | 3.33 [1.2 to 7.0] | 3.37 [1.2 to 7.0] | 3.53 [1.3 to 6.7] | 3.29 [1.2 to 7.6]
  Week 4 change from Baseline: number analyzed (Participants) | 207 | 103 | 105 | 203
  Week 4 change from Baseline | -2.64 [-6.1 to 1.8] | -2.76 [-6.9 to 0.9] | -2.48 [-4.9 to 1.6] | -2.81 [-6.1 to 1.8]
  Week 8: number analyzed (Participants) | 202 | 103 | 104 | 204
  Week 8 | 3.28 [1.2 to 7.2] | 3.37 [1.2 to 6.9] | 3.51 [1.2 to 6.6] | 3.25 [1.2 to 7.1]
  Week 8 change from Baseline: number analyzed (Participants) | 201 | 102 | 104 | 204
  Week 8 change from Baseline | -2.72 [-5.9 to 2.7] | -2.74 [-6.9 to 0.8] | -2.47 [-4.8 to 0.9] | -2.84 [-5.8 to -0.2]
  Week 12: number analyzed (Participants) | 200 | 102 | 103 | 203
  Week 12 | 3.31 [1.2 to 6.9] | 3.30 [1.2 to 7.1] | 3.40 [1.3 to 6.2] | 3.21 [1.2 to 6.5]
  Week 12 change from Baseline: number analyzed (Participants) | 199 | 101 | 103 | 203
  Week 12 change from Baseline | -2.70 [-5.9 to 0.8] | -2.80 [-6.9 to 0.3] | -2.57 [-4.9 to 0.5] | -2.88 [-5.8 to 0.9]
  Week 24: number analyzed (Participants) | 197 | 98 | 95 | 197
  Week 24 | 3.13 [1.2 to 7.8] | 3.27 [1.2 to 7.1] | 3.40 [1.2 to 7.7] | 3.07 [1.2 to 7.5]
  Week 24 change from Baseline: number analyzed (Participants) | 196 | 97 | 95 | 197
  Week 24 change from Baseline | -2.89 [-6.1 to 1.3] | -2.86 [-6.7 to 0.9] | -2.57 [-5.4 to 1.7] | -3.04 [-6.0 to -0.0]
  Period II: Week 30: number analyzed (Participants) | 183 | 99 | 92 | 189
  Period II: Week 30 | 3.04 [1.2 to 7.1] | 3.28 [1.2 to 7.1] | 3.20 [1.3 to 6.3] | 3.13 [1.2 to 7.4]
  Week 30 change from Baseline: number analyzed (Participants) | 182 | 98 | 92 | 189
  Week 30 change from Baseline | -2.99 [-6.1 to 0.3] | -2.84 [-6.6 to 0.5] | -2.78 [-5.3 to 0.4] | -2.95 [-6.2 to 1.9]
  Week 42: number analyzed (Participants) | 184 | 96 | 90 | 187
  Week 42 | 3.05 [1.2 to 6.8] | 3.28 [1.2 to 6.1] | 3.08 [1.3 to 6.0] | 3.07 [1.2 to 7.3]
  week 42 change from Baseline: number analyzed (Participants) | 183 | 95 | 90 | 187
  week 42 change from Baseline | -2.97 [-5.6 to 0.9] | -2.83 [-6.2 to -0.2] | -2.88 [-5.5 to -0.0] | -3.01 [-5.8 to 0.6]
  Week 54: number analyzed (Participants) | 180 | 92 | 89 | 180
  Week 54 | 3.04 [1.2 to 7.5] | 3.22 [1.2 to 6.2] | 3.26 [1.2 to 6.2] | 2.96 [1.2 to 6.8]
  Week 54 change from Baseline: number analyzed (Participants) | 179 | 91 | 89 | 180
  Week 54 change from Baseline | -2.99 [-5.9 to 0.4] | -2.90 [-6.2 to 0.9] | -2.70 [-5.4 to 0.4] | -3.12 [-5.6 to 1.6]
  Week 66: number analyzed (Participants) | 174 | 89 | 84 | 175
  Week 66 | 2.96 [1.2 to 7.0] | 3.17 [1.2 to 5.7] | 3.09 [1.3 to 5.6] | 2.91 [1.2 to 6.9]
  Week 66 change from Baseline: number analyzed (Participants) | 173 | 88 | 84 | 175
  Week 66 change from Baseline | -3.09 [-5.9 to 0.3] | -2.96 [-6.9 to -0.0] | -2.83 [-5.5 to 0.8] | -3.15 [-5.6 to 0.2]
  Week 76: number analyzed (Participants) | 174 | 90 | 81 | 172
  Week 76 | 2.97 [1.2 to 7.8] | 3.02 [1.2 to 6.2] | 3.12 [1.3 to 7.0] | 2.94 [1.2 to 6.4]
  Week 76 change from Baseline: number analyzed (Participants) | 173 | 89 | 81 | 172
  Week 76 change from Baseline | -3.04 [-5.9 to 0.2] | -3.11 [-6.1 to 0.4] | -2.79 [-5.5 to 1.0] | -3.14 [-5.7 to -0.2]
  Week 80: number analyzed (Participants) | 172 | 88 | 81 | 170
  Week 80 | 2.98 [1.2 to 7.1] | 3.09 [1.2 to 6.9] | 3.25 [1.2 to 6.7] | 3.06 [1.2 to 6.7]
  Week 80 change from Baseline: number analyzed (Participants) | 171 | 87 | 81 | 170
  Week 80 change from Baseline | -3.05 [-6.2 to 2.2] | -3.05 [-6.9 to -0.3] | -2.66 [-5.4 to 0.2] | -3.02 [-5.8 to 0.2]

11. Secondary Outcome: American College of Rheumatology 20 (ACR20) Response Rates From Baseline as a Measure of Efficacy
Description: An ACR20 response means that the patient achieved a 20% improvement in Tender Joint Count (TJC) and Swollen Joint Count (SJC) and a 20% improvement in at least 3 of the other 5 Core Data Set elements listed below:
  * Acute phase reactant (C-reactive protein, CRP) A high level of CRP in the blood is a marker of inflammation.
  * Patient global assessment of disease activity assessed on a Visual Analog Scale (VAS) ranging from very well to extremely bad was assessed on a 100 point scale. (from 0 to 100)
  * Physician global assessment of disease activity assessed on a VAS ranging from very low to very high was assessed on 100 point scale
  * Patient pain scale assessed on a VAS ranging from very well to extremely bad was assessed on 100 point scale
  * Disability/functional questionnaire (patient completed Heath Assessment Questionnaire Disability Index (HAQ-DI)) A higher response rate is a better outcome. The minimum possible value is 0% and the maximum possible value is 100%
Time Frame: From Week 0 to Week 80
Population: Number of patients at a given time-point with an observed ACR20 score defined as a 20% improvement in tender and swollen joints and at least 3 out of 5 other indicators from Baseline_002 (Week 0 of FKB327-002; NCT02260791)
Measure: Count of Participants; unit: Participants
Groups:
- FKB327-FKB327-FKB327: Period I: This is the treatment arm where subjects had been treated with FKB327 in the preceding study, FKB327-002 and were re-randomized to FKB327 in Period I of study FKB327-003 (F-F).
  Period II: From week 30 all subjects received FKB327 (F-F-F).
- FKB327-Humira-FKB327: Period I: This is the treatment arm where subjects had been treated with FKB327 in the preceding study FKB327-002 and were re-randomized to the reference product, Humira, during Period I of study FKB327-003 (F-H).
  Period II: From week 30 all subjects received FKB327 (F-H-F).
- Humira-FKB327-FKB327: Period I: This is the treatment arm where subjects had been treated with the reference product Humira in the preceding study, FKB327-002 and were re-randomized to FKB327 during Period I of study FKB327-003 (H-F).
  Period II: From week 30 all subjects received FKB327 (H-F-F).
- Humira-Humira-FKB327: Period I: This is the treatment arm where subjects had been treated with the reference product Humira in the preceding study, FKB327-002, and were re-randomized to the reference product Humira during Period I of study FKB327-003 (H-H).
  Period II: From week 30 all subjects received FKB327 (H-H-F).
Arm/Group | FKB327-FKB327-FKB327 | FKB327-Humira-FKB327 | Humira-FKB327-FKB327 | Humira-Humira-FKB327
Number analyzed (Participants) | 216 | 108 | 108 | 213
Participants
  Week 0: number analyzed (Participants) | 216 | 108 | 108 | 212
  Week 0 | 163 | 87 | 82 | 175
  Week 4: number analyzed (Participants) | 210 | 105 | 107 | 208
  Week 4 | 171 | 83 | 84 | 165
  Week 8: number analyzed (Participants) | 205 | 103 | 104 | 204
  Week 8 | 160 | 84 | 79 | 173
  Week 12: number analyzed (Participants) | 203 | 102 | 103 | 203
  Week 12 | 160 | 89 | 82 | 171
  Week 24: number analyzed (Participants) | 197 | 100 | 95 | 198
  Week 24 | 162 | 83 | 75 | 176
  Period II: Week 30: number analyzed (Participants) | 185 | 98 | 92 | 189
  Period II: Week 30 | 154 | 82 | 79 | 158
  Week 42: number analyzed (Participants) | 184 | 96 | 90 | 187
  Week 42 | 156 | 79 | 81 | 164
  Week 54: number analyzed (Participants) | 180 | 93 | 90 | 180
  Week 54 | 149 | 78 | 77 | 152
  Week 66: number analyzed (Participants) | 174 | 89 | 84 | 175
  Week 66 | 140 | 73 | 74 | 150
  Week 76: number analyzed (Participants) | 175 | 90 | 81 | 172
  Week 76 | 140 | 77 | 71 | 147
  Week 80/EOS: number analyzed (Participants) | 173 | 88 | 81 | 170
  Week 80/EOS | 133 | 72 | 62 | 140

12. Secondary Outcome: American College of Rheumatology 50 (ACR50) Response Rates From Baseline as a Measure of Efficacy
Description: An ACR50 response means that the patient achieved a 50% improvement in Tender Joint Count (TJC) and Swollen Joint Count (SJC) and in at least 3 of the other 5 Core Data Set elements listed below:
  * Acute phase reactant (C-reactive protein, CRP) A high level of CRP in the blood is a marker of inflammation.
  * Patient global assessment of disease activity assessed on a Visual Analog Scale (VAS) ranging from very well to extremely bad was assessed on a 100 point scale. (from 0 to 100)
  * Physician global assessment of disease activity assessed on a VAS ranging from very low to very high was assessed on 100 point scale
  * Patient pain scale assessed on a VAS ranging from very well to extremely bad was assessed on 100 point scale
  * Disability/functional questionnaire (patient completed Heath Assessment Questionnaire Disability Index (HAQ-DI)) A higher response rate is a better outcome. The minimum possible value is 0% and the maximum possible value is 100%
Time Frame: From Week 0 to Week 80
Population: Number of patients at a given time-point with an observed ACR50 score defined as a 50% improvement in tender and swollen joints and at least in 3 out of 5 other indicators from Baseline_002 (Week 0 of FKB327-002; NCT02260791)
Measure: Count of Participants; unit: Participants
Arm/Group | FKB327-FKB327-FKB327 | FKB327-Humira-FKB327 | Humira-FKB327-FKB327 | Humira-Humira-FKB327
Number analyzed (Participants) | 216 | 108 | 108 | 213
Participants
  Week 0: number analyzed (Participants) | 215 | 108 | 108 | 212
  Week 0 | 104 | 52 | 50 | 109
  Week 4: number analyzed (Participants) | 211 | 105 | 107 | 208
  Week 4 | 110 | 50 | 52 | 115
  Week 8: number analyzed (Participants) | 205 | 103 | 104 | 204
  Week 8 | 106 | 53 | 51 | 124
  Week 12: number analyzed (Participants) | 202 | 102 | 103 | 203
  Week 12 | 106 | 53 | 55 | 131
  Week 24: number analyzed (Participants) | 197 | 100 | 95 | 199
  Week 24 | 114 | 56 | 49 | 127
  Period II: Week 30: number analyzed (Participants) | 185 | 98 | 92 | 189
  Period II: Week 30 | 112 | 57 | 50 | 113
  Week 42: number analyzed (Participants) | 184 | 96 | 90 | 187
  Week 42 | 113 | 47 | 54 | 115
  Week 54: number analyzed (Participants) | 180 | 92 | 90 | 180
  Week 54 | 106 | 47 | 44 | 110
  Week 66: number analyzed (Participants) | 174 | 89 | 84 | 175
  Week 66 | 110 | 48 | 46 | 114
  Week 76: number analyzed (Participants) | 175 | 90 | 81 | 173
  Week 76 | 108 | 59 | 43 | 108
  Week 80/EOS: number analyzed (Participants) | 173 | 88 | 81 | 170
  Week 80/EOS | 102 | 47 | 43 | 112

13. Secondary Outcome: American College of Rheumatology 70 (ACR70) Response Rates From Baseline as a Measure of Efficacy
Description: An ACR70 response means that the patient achieved a 70% improvement in Tender Joint Count (TJC) and Swollen Joint Count (SJC) and in at least 3 of the other 5 Core Data Set elements listed below:
  * Acute phase reactant (C-reactive protein,CRP) A high level of CRP in the blood is a marker of inflammation.
  * Patient global assessment of disease activity assessed on a Visual Analog Scale (VAS) ranging from very well to extremely bad was assessed on a 100 point scale. (from 0 to 100)
  * Physician global assessment of disease activity assessed on a VAS ranging from very low to very high was assessed on 100 point scale
  * Patient pain scale assessed on a VAS ranging from very well to extremely bad was assessed on 100 point scale
  * Disability/functional questionnaire (patient completed Heath Assessment Questionnaire Disability Index (HAQ-DI)) A higher response rate is a better outcome. The minimum possible value is 0% and the maximum possible value is 100%
Time Frame: From Week 0 to Week 80
Population: Number of patients at a given time-point with an observed ACR70 score defined as a 70% improvement in tender and swollen joints and at least 3 out of 5 other indicators from Baseline_002 (Week 0 of FKB327-002; NCT02260791)
Measure: Count of Participants; unit: Participants
Arm/Group | FKB327-FKB327-FKB327 | FKB327-Humira-FKB327 | Humira-FKB327-FKB327 | Humira-Humira-FKB327
Number analyzed (Participants) | 216 | 108 | 108 | 213
Participants
  Week 0: number analyzed (Participants) | 216 | 108 | 108 | 212
  Week 0 | 45 | 23 | 23 | 56
  Week 4: number analyzed (Participants) | 211 | 104 | 107 | 207
  Week 4 | 54 | 30 | 29 | 54
  Week 8: number analyzed (Participants) | 204 | 103 | 104 | 204
  Week 8 | 61 | 29 | 26 | 72
  Week 12: number analyzed (Participants) | 203 | 102 | 103 | 203
  Week 12 | 59 | 28 | 29 | 69
  Week 24: number analyzed (Participants) | 197 | 99 | 95 | 199
  Week 24 | 65 | 30 | 25 | 80
  Period II: Week 30: number analyzed (Participants) | 185 | 99 | 92 | 189
  Period II: Week 30 | 67 | 33 | 28 | 74
  Week 42: number analyzed (Participants) | 184 | 96 | 90 | 187
  Week 42 | 72 | 27 | 26 | 74
  Week 54: number analyzed (Participants) | 180 | 93 | 90 | 180
  Week 54 | 69 | 29 | 19 | 69
  Week 66: number analyzed (Participants) | 174 | 89 | 84 | 175
  Week 66 | 69 | 29 | 25 | 73
  Week 76: number analyzed (Participants) | 175 | 90 | 81 | 173
  Week 76 | 72 | 31 | 20 | 71
  Week 80/EOS: number analyzed (Participants) | 172 | 88 | 81 | 170
  Week 80/EOS | 64 | 27 | 25 | 69

14. Other Pre Specified Outcome: Proportion of Patients Developing Anti-drug Antibodies (ADAs)
Description: Blood samples for assessment of Anti-Drug antibodies (ADA) were collected prior to dosing (trough samples) at Baseline (Week 0) and at Weeks 12, 24, 30, 54, 76 and 80/EOS.
  All ADA activity was listed and summarized for each treatment sequence by time point during the overall treatment period as well as by treatment group for each period (Period I and Period II). Descriptive statistics included absolute counts (n) and percentage (%).
Time Frame: From Week 0 to Week 80
Population: Number of patients who had an assay result of positive Anti-Drug Antibodies at given time-points.
Measure: Count of Participants; unit: Participants
Groups:
- FKB327-Humira-FKB327: Period I: This is the treatment arm where subjects had been treated with FKB327 in the preceding study FKB327-002 and were re-randomized to the reference product Humira during Period I of study FKB327-003 (F-H).
  Period II: From week 30 all subjects received FKB327 (F-H-F).
Arm/Group | FKB327-FKB327-FKB327 | FKB327-Humira-FKB327 | Humira-FKB327-FKB327 | Humira-Humira-FKB327
Number analyzed (Participants) | 216 | 108 | 108 | 213
Participants
  Week 0: number analyzed (Participants) | 216 | 108 | 108 | 212
  Week 0 | 133 | 69 | 67 | 123
  Week 12: number analyzed (Participants) | 202 | 103 | 103 | 202
  Week 12 | 107 | 60 | 54 | 101
  Week 24: number analyzed (Participants) | 197 | 100 | 96 | 199
  Week 24 | 99 | 58 | 47 | 100
  Period II: Week 30: number analyzed (Participants) | 187 | 100 | 93 | 190
  Period II: Week 30 | 97 | 61 | 42 | 98
  Week 54: number analyzed (Participants) | 181 | 93 | 89 | 181
  Week 54 | 103 | 49 | 41 | 77
  Week 76: number analyzed (Participants) | 176 | 90 | 81 | 174
  Week 76 | 90 | 49 | 39 | 74
  Week 80/EOS: number analyzed (Participants) | 173 | 87 | 80 | 170
  Week 80/EOS | 91 | 48 | 37 | 72
  Last Sampling Day | 115 | 63 | 49 | 99

15. Other Pre Specified Outcome: Trough Adalimumab Concentration
Description: Blood samples for the quantification of adalimumab concentration in serum were collected prior to dosing (trough samples) at Baseline (Week 0), and at weeks 12, 24 , 30, 54, 76 and 80/EOS.
Time Frame: From Week 0 to Week 80
Population: Analysis of Serum Concentration Data (ng/mL). Repeated measure of pharmacokinetic(s) (PK) trough concentrations at given time-points.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Humira-Humira-FKB327: Period I: This is the treatment arm where subjects had been treated with the reference product Humira in the preceding study, FKB327-002, and were re-randomized to the reference product Humira during Period I of study FKB327-003 (H-H).
  Period I: From week 30 all subjects received FKB327 (H-H-F).
Arm/Group | FKB327-FKB327-FKB327 | FKB327-Humira-FKB327 | Humira-FKB327-FKB327 | Humira-Humira-FKB327
Number analyzed (Participants) | 208 | 105 | 107 | 210
ng/mL
  Week 0: number analyzed (Participants) | 208 | 105 | 107 | 209
  Week 0 | 6500 (4640) | 6000 (4520) | 5170 (3440) | 5720 (3470)
  Week 12: number analyzed (Participants) | 202 | 103 | 103 | 202
  Week 12 | 6310 (4720) | 5380 (4150) | 6180 (3970) | 6010 (3730)
  Week 24: number analyzed (Participants) | 197 | 100 | 95 | 199
  Week 24 | 5970 (4500) | 5100 (3990) | 6320 (4320) | 5950 (3750)
  Period II: Week 30: number analyzed (Participants) | 187 | 100 | 93 | 190
  Period II: Week 30 | 6000 (4450) | 4790 (4290) | 5730 (3750) | 5750 (3680)
  Week 54: number analyzed (Participants) | 180 | 93 | 89 | 181
  Week 54 | 6090 (4620) | 5830 (4290) | 5840 (4100) | 6620 (3920)
  Week 76: number analyzed (Participants) | 176 | 90 | 80 | 173
  Week 76 | 6460 (4140) | 5900 (4020) | 6070 (4350) | 6730 (4080)
  Week 80: number analyzed (Participants) | 173 | 87 | 80 | 170
  Week 80 | 4320 (3130) | 4000 (3280) | 4060 (3310) | 4520 (3100)

ADVERSE EVENTS:
Time Frame: Overall Adverse Events and Serious Adverse Events were collected and monitored up to week 80 for subjects completing the study and 4 weeks after an Early Termination Visit. Period I - from signing of informed consent up to week 30. During this period subjects received either FKB327 or the reference product Humira. Period II: From week 30 to week 76 all subjects received FKB327 hence the maximum duration of FKB327 treatment was about 2.5 times greater compared to the Humira (581 vs 222 days).
Description: The overall exposure in patient-years was nearly 4 times greater for FKB327 (673.7) compared to Humira (175.4), due to patients switching from Humira to FKB327 for Period II, which should be taken into account when reviewing the safety results where FKB327 and Humira are directly compared.
Groups:
- FKB327: FKB327: Solution of FKB327 for subcutaneous injection administered in a dose of 40 mg/0.8mL every 2 weeks for 28 weeks. From week 30 all patients were transferred to receive FKB327 40 mg/0.8 mL every other week presented in an auto-injector (AI) or a pre-filled syringe (PFS). Some patients received continuous FKB327 40 mg every other week by subcutaneous injection for up to 76 weeks.
- Humira®: Humira®: Solution of Humira® for subcutaneous injection administered in a dose of 40 mg every 2 weeks for 28 weeks. From week 30 to week 76 all patients were transferred to receive FKB327 40 mg/0.8 mL in a pre-filled syringe (PFS) every other week by subcutaneous injection.
Arm/Group | FKB327 | Humira®
All-Cause Mortality (participants affected / at risk) | 3/614 | 1/321
Serious Adverse Events (participants affected / at risk) | 43/614 | 14/321
Other Adverse Events (participants affected / at risk) | 125/614 | 46/321
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FKB327 (N=614) | Humira® (N=321)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (2)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Oesophageal rupture (Gastrointestinal disorders) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Sudden death (General disorders) | 1 (1) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis chronic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatocellular injury (Hepatobiliary disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 4 (4) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 4 (4) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1)
Pyelonephritis (Infections and infestations) | 2 (2) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0)
Meningitis (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary mycosis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Maternal exposure during pregnancy (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Muscle rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Back disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Synovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Anterior spinal artery syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure chronic (Renal and urinary disorders) | 0 (0) | 1 (1)
Cervical dysplasia (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hip arthroplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
Joint surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
Knee Arthroplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Synovectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Lymphostatis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FKB327 (N=614) | Humira® (N=321)
Nasopharyngitis (Infections and infestations) | 68 (77) | 22 (25)
Bronchitis (Infections and infestations) | 32 (34) | 14 (15)
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 37 (53) | 15 (18)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator and Sponsor will discuss the preparation of a manuscript for publication in a peer reviewed journal or an abstract for presentation. Either party may undertake the task but both must agree to the strategy before work is started. Each party will allow the other 30 days to comment before any results are submitted for publication or presentation. Authorship should reflect work done by the Investigator an Sponsor, in accordance with recognized principles of scientific collaboration.

DOCUMENTS (2):
  • Study Protocol (2016-04-15): https://cdn.clinicaltrials.gov/large-docs/80/NCT02405780/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-10): https://cdn.clinicaltrials.gov/large-docs/80/NCT02405780/SAP_001.pdf